CLINICAL TRIAL: NCT06679634
Title: Retinoblastoma Phase II Expanded Access Clinical Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Targeted Therapy Technologies, LLC (Industry)
Collaborators: Morgan Stanley Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3TRB01-2
Record Dates: First submitted 2024-11-05; First posted 2024-11-07 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Retinoblastoma
Keywords: Retinoblastoma
MeSH Terms: conditions — Retinoblastoma

STUDY DESIGN:
Intervention Model Description: Single Arm Open Label Expanded Access
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Chemoplaque (Experimental): Chemoplaque (also referred to as Episcleral Topotecan) treatment will involve single application of the Episcleral Topotecan 1.2 mg dose that delivers sustained delivery for 8 weeks.
  Interventions: Drug: Chemoplaque also referred to as Episcleral Topotecan

INTERVENTIONS:
Drug: Chemoplaque also referred to as Episcleral Topotecan — Sustained Release Episcleral Topotecan
  Other Names: Episcleral Topotecan

SUMMARY:
In this research study investigators want to learn more about treatment of advanced or recurrent retinoblastoma. For children with retinoblastoma that have an advanced stage of presentation in one eye or if they have failed all conventional treatment, eye removal is considered. This study will investigate the utility of a chemoplaque(s) to salvage eyes involved with retinoblastoma. The goal of the study is to further determine/assess the safety and efficacy and optimal chemotherapy dose for retinoblastoma.

DETAILED DESCRIPTION:
The chemoplaque will be placed during the first exam under anesthesia (EUA) and this involves a surgery wherein the reservoir that will release the chemotherapy medication will be placed under the conjunctiva (surface lining of the eye) and will be applied with tissue adhesive to the sclera (coating of the eye). The chemoplaque will remain on the eye until day 56 when the chemoplaque will be removed. Eye exam under anesthesia (EUAs) will be performed on Day 0, Day 28, Day 56 (prior to chemoplaque removal), and Day 84 (final visit). Blood will be drawn periodically for testing the blood parameters (CBC) and to evaluate toxicity of the medication. Study subjects will be followed until Day 84 when protocol therapy will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Age: Participants must be < 8 years of age.
* Diagnosis and Treatment. Participants must have: Group D or earlier-stage intraocular retinoblastoma in which enucleation is a recommended therapy, OR Active residual or recurrent intraocular retinoblastoma in at least one eye following completion of first- line therapy (focal therapy for IIRC Group A eyes, or systemic or intra-arterial chemotherapy).

If both eyes require treatment, there will receive independent and individual treatment. Non-study eye will be treated by standard of care, with only focal therapy during the Study Period, if required.

* Must have demonstrated intraocular calcium in the tumor-containing eye by ophthalmic ultrasound or by neuroimaging as part of standard retinoblastoma diagnosis.
* Study eye must have vision potential, at least light perception vision in the tumor-bearing eye either with pupil response testing or demonstration of avoidance behavior to light presentation in the affected eye, and no clinical features suggestive of high risk of extraocular extension.
* Performance Level: Lansky ≥ 50 (<16 years of age); Karnofsky performance scale of ≥50 (≥16 years of age).
* Organ Function Requirements:

  1. Adequate Bone Marrow Function defined as:

     * Peripheral absolute neutrophil count (ANC) ≥ 1000/mm3
     * Platelet count ≥ 100,000/mm3 (transfusion independent, defined as not receiving platelet transfusions for at least 7 Days prior to enrollment)
     * Hemoglobin ≥ 8.0 g/dL at baseline (may receive RBC transfusions)
  2. Adequate Renal Function defined as:

     * Creatinine clearance or radioisotope GFR ≥70ml/min/1.73 m2 or
     * A serum creatinine based on age/gender as follows:

     Age Maximum Serum Creatinine (mg/dL) Male Female

     1 month to < 6 months 0.4 0.4 6 months to < 1 year 0.5 0.5
     1. to < 2 years 0.6 0.6
     2. to < 6 years 0.8 0.8

     6 to < 7 years 1 1

     The threshold creatinine values in this Table were derived from the Schwartz formula for estimating GFR utilizing child length and stature data published by the CDC.
  3. Adequate Liver Function defined as:

     * Bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x upper limit of normal (ULN) for age.
     * SGPT (ALT) ≤ 110 U/L. For the purpose of this study, the ULN for SGPT is 45 U/L.
     * Serum albumin ≥ 2 g/dL.
  4. Pregnancy prevention. Females of reproductive potential must agree to the use of highly effective contraception during study participation and for an additional 40 days after the end of Episcleral Topotecan administration.
  5. Informed consent. All participants and/or their parents or legally authorized representatives must have the ability to understand and the willingness to sign a written informed consent. Assent, where appropriate, will also be obtained.

Exclusion Criteria:

* Disease status. Participants known to have any of the following are excluded:

  1. tumor involving the optic nerve rim
  2. clinical or EUA evidence of extraocular extension
  3. evidence of metastatic retinoblastoma
  4. existing neuroimaging showing suspicion of, or definitive, optic nerve invasion, trilateral retinoblastoma or extra-ocular extension.
* Allergy. Participants with reported allergy to topotecan, camptothecin or derivatives thereof are excluded.
* Concomitant treatment. Participants who have received chemotherapy, other focal retinoblastoma therapy or any other investigational agent within 3 weeks of Episcleral Topotecan placement are not eligible.
* Uncontrolled intercurrent illness. Participants with known uncontrolled intercurrent illness that, in the investigator's opinion, would put the participant at undue risk or limit compliance with the study requirements, are not eligible.
* Febrile illness. Participants with clinically significant febrile illness (as determined by the investigator) within one week prior to initiation of protocol therapy are excluded.
* Pregnancy and lactation. Females of reproductive potential must have a negative serum pregnancy test within 72 hours prior to initiation of protocol therapy. Due to the unknown but potential risk for adverse events (AEs) in nursing infants secondary to treatment of the mother with the study agents, breastfeeding must be discontinued if the mother is treated on study.
* Compliance. Any condition of diagnosis that could in the opinion of the Principal Investigator or delegate interfere with the participant's ability to comply with the study instruction, might confound the interpretation of the study results, or put the participant at risk.

Max Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
To determine the safety and tolerability of Episcleral Topotecan in participants with retinoblastoma by measuring the rate and severity of treatment related adverse events in study participants as assessed by CTCAE version 5.0 criteria. | 12 weeks and follow up

SECONDARY OUTCOMES:
To determine the safety and tolerability of Episcleral Topotecan in participants with retinoblastoma by measuring the rate and severity of treatment related ocular adverse events in study participants as assessed by CTCAE version 5.0 criteria. | 12 weeks and follow up
To determine the safety and tolerability of Episcleral Topotecan in participants with retinoblastoma by measuring the rate and severity of treatment related systemic adverse events in study participants as assessed by CTCAE version 5.0 criteria. | 12 weeks
To describe the anti-tumor efficacy of Episcleral Topotecan | 12 weeks and follow up
  Tumor response will be assessed via image analysis with following criteria: Complete Response (CR): Decrease in tumor activity 100% from baseline. Very good partial response (VGPR): Decrease in tumor activity greater than or equal to 80% and less than 100% from baseline. Partial response (PR): Decrease in tumor activity greater than or equal to 20% and less than 80% from baseline. Stable disease (SD): Less than 20% decrease in tumor activity from baseline. Progressive disease (PD): Increase in tumor activity greater than or equal to 20% from baseline or development of new tumours requiring more than minimal focal therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- NewYork Presbyterian Morgan Stanley Children's Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No